CLINICAL TRIAL: NCT04386538
Title: Effect of a Low Starch Diet in the Gut Microbiome Modulation, Disease Activity and Quality of Life in Patients With Ankylosing Spondylitis
Brief Title: Effect of a Low Starch Diet in Patients With Ankylosing Spondylitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Portuguese Institute of Rheumatology (Unknown); Centro de Investigação Interdisciplinar Egas Moniz (Unknown)
Responsible Party: Principal Investigator, Alexandra Cardoso, Principal investigator, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: alexandracardoso
Record Dates: First submitted 2020-05-04; First posted 2020-05-13 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Spondyloarthritis; Ankylosing Spondylitis
Keywords: Low Starch Diet (LSD); Klebsiella; Ankylosing Spondylitis; Disease activity; Quality of life; Nutrition; Diet therapy; Spondyloarthritis; Rheumatic Diseases; Spondylitis
MeSH Terms: conditions — Spondylarthritis; Spondylitis, Ankylosing; Klebsiella Infections; Rheumatic Diseases; Spondylitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Starch Diet (LSD) (Experimental): Participants will receive the low starch diet program: restricts the daily amount of ingested rich starch food, to a reduction of at least 40% compared to usual daily individual starch intake.
  Interventions: Behavioral: Low Starch Diet (LSD)
- Control (Active Comparator): Participants will receive dietary counselling based on general recommendations for healthy eating.
  Interventions: Behavioral: General healthy eating

INTERVENTIONS:
Behavioral: Low Starch Diet (LSD) — 6-week balanced diet program, adapted to individual energetic needs, with significant reduction of high content starchy food, naturally present in plant cells, roots, tubers, seeds, beans, legumes, fruits, and highly present in most farinaceous grains, especially in potatoes, corn, rice, pasta, bread, cookies and cakes.
  Arms: Low Starch Diet (LSD)
Behavioral: General healthy eating — 6-week balanced healthy eating counseling program, according to the World Health Organization recommendations.
  Arms: Control

SUMMARY:
The aim of this study is to explore the effect of a low starch diet (reduction of at least 40%) in the gut bacteria modulation, especially Klebsiella pneumoniae, and its relation to disease activity, functional impairment and quality of life in patients with Ankylosing Spondylitis (AS).

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is a chronic inflammatory rheumatic disease characterized by axial inflammation and with unknown aetiology. The immune system dysregulation is known, where genetic factors play a key role, in particular, the susceptibility associated to the HLA-B27 allele. The presence of this genetic marker, seems to trigger an abnormal response of the individual, under the action of determine microorganisms, and probably, the combination of these two factors may contribute to the manifestation of the disease, through the induction of an immune and cytolytic response, leading to tissue injury and promoting the inflammation. Intestinal microbiota involvement in spondylarthritis is a controversial issue, however, was observed an increased concentration of Klebsiella pneumoniae bacteria in the faeces of AS patients. It has been suggested that an intervention aiming these bacteria's starving could benefit the reduction of the inflammatory processes and be a part of AS treatment. The bowel microflora depends on dietary intake, like undigested starch, for their growth. Some studies have highlighted the relation between the intake of starch and the disease activity. The modulation of the microbiota, particularly, the reduction of Klebsiella, may be beneficial as a complementary approach to AS therapy.

A sample of 300 patients with AS, followed-up at Portuguese Institute of Rheumatology in Lisbon, will be randomly assigned in two groups. The group A will adopt a balanced diet based on the general recommendations for healthy eating by the World Health Organization, for a period of 6 weeks. In Group B will be implemented an individual balanced low starch diet, which is characterized by the significant reduction of starchy food, of at least 40% of the total daily ingested starch.

The change in biometric data, body composition, intestinal Klebsiella will be related to food intake, disease activity and quality of life assessments. These data will be compared between the 2 groups (diet A versus diet B), obtaining measures on the effect of each diet on the analyzed variables.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years old
* Available to comply with study protocol
* Ability to read and sign the Informed Consent
* Diagnosis of Ankylosing Spondylitis performed by the rheumatologist, according to the ASAS classification criteria, revised in 2016
* Positive HLA-B27allele
* Stable dose therapy within 3 months before selection

Exclusion Criteria:

* Pregnant, breastfeeding or planning to become pregnant within the study period
* Prior or current clinical history of drug or other substances abuse
* Subjects with uncontrolled clinical conditions, like neoplastic diseases, renal failure, liver impairment, uncompensated cardiac disease
* Dietetic restrictions due to religious believes or others incompatible with the study protocol
* Impossibility to attend to the mandatory personal clinical evaluation
* Presence of pacemaker, making impossible to perform the impedance body composition analysis
* Change in therapy during the intervention period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in intestinal Klebsiella | 6 weeks (at baseline and the end of follow-up between the two groups)
  To compare the mean change of Klebsiella bacteria in faecal samples between the LSD group and the control.
Change in mean erythrocyte sedimentation rate (ESR) | 6 weeks (at baseline and the end of follow-up)
  Plasma concentrations will be assessed to evaluate ESR, a marker of systemic inflammation that provided insights into the overall anti-inflammatory effect of rheumatologic therapies. Data are presented as mean ESR value in millimeters per hour (mm/hr) ± standard deviation.
Change in mean C-reactive protein (CRP) | 6 weeks (at baseline and the end of follow-up)
  Plasma concentrations will be assessed to evaluate CRP, a marker of systemic inflammation that provided insights into the overall anti-inflammatory effect of rheumatologic therapies. Data are presented as mean CRP value in milligrams per liter (mg/L) ± standard deviation.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 6 weeks (at baseline and the end of follow-up)
  The BASDAI is a six question, participant-reported measure of overall disease activity that probed the level of fatigue, neck/back/hip pain, peripheral joint swelling and pain, localized tenderness, as well as morning stiffness severity and duration. The mean measurement (score) of questions 5 and 6 is added to the scores from questions 1 to 4 and divided by 5 to calculate the total BASDAI score. It is scored on a numerical rating scale that ranges from 0 (no symptoms) to 10 (severe symptoms), higher scores indicating severe disability due to AS disease. Data are presented as mean total BASDAI score +/- standard deviation.
Bath Ankylosing Spondylitis Function Index (BASFI) | 6 weeks (at baseline and the end of follow-up)
  The BASFI is a self-assessment instrument used to assess function. It comprises 8 specific questions regarding function in AS and 2 questions to identify participant's ability to cope up with everyday life. Each question is answered on a 100 millimeter (mm) horizontal VAS. The mean VAS score gives BASFI score between 0 to 100 where 0=easy to 100=impossible.
Ankylosing Spondylitis Disease Activity Score (ASDAS) | 6 weeks (at baseline and the end of follow-up)
  ASDAS includes CRP mg/L; four additional self-reported items (rated on 0-10cm VAS or 0-10 numerical rating scale [NRS]) included are total back pain (TBP), duration of morning stiffness (DMS), peripheral pain/swelling and patient global assessment (PGA). ASDAS scores calculated as: ASDAS(CRP) = (0.121*total back pain) + (0.110*participant global) + (0.073*peripheral pain/swelling) + (0.058* duration of morning stiffness) + (0.579*Ln(CRP+1). The disease activity, TBP, and peripheral pain/swelling on a numeric rating scale (from 0 (normal) to 10 (very severe)) and DMS on a numeric rating scale (0 to 10, with 0 being none and 10 representing a duration of =>2 hours). Inactive disease is defined as an ASDAS score <1.3.
Bath Ankylosing Spondylitis Patient Global Score (BAS-G) | 6 weeks (at baseline and the end of follow-up)
  The self-administered Bath Ankylosing Spondylitis Global (BAS-G) measures global consequences of axial spondyloarthritis, indicating the effect of disease on participant's well-being. This scale is composed of 2 items ranging from 0 = very good to 10 =very bad. Total score ranges from 0 to 10: the higher the BAS-G score, the worse the participant's health status.
Ankylosing Spondylitis Quality of Life (ASQoL) | 6 weeks (at baseline and the end of follow-up)
  The Ankylosing Spondylitis Quality of Life (ASQoL) questionnaire is a disease-specific instrument designed to measure the health related quality of life (HRQOL) in participants with AS. Participants answer yes/no to 18 items assessing the current impact of AS on their quality of life status. The total score ranges from 0 to 18, with lower scores representing better AS-specific quality of life. Negative numbers indicate improvement from baseline.
Euro Quality of Life-5D (EQ-5D) | 6 weeks (at baseline, 2-weeks, 4-weeks, end of follow-up)
  The EQ-5D is a standardized, generic measure of health outcome, designed for self-completion by participants. The EQ-5D includes a descriptive section with 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) that are combined into an overall health utilities index, and an NRS (100 mm VAS) that measures perception of overall health, with 0 indicating worst health and 100 representing best imaginable health.
Change in Short Form (36) Health Survey (SF-36) | 6 weeks (at baseline and the end of follow-up)
  SF-36 is a generic 36-item questionnaire measuring health-related quality of life (HRQL) covering 2 summary measures: physical component summary (PCS) and mental component summary (MCS). The SF-36 consists of 8 subscales. The PCS had 4 subscales: physical function, role limitations due to physical problems, pain, and general health perception. The MCS had 4 subscales: vitality, social function, role limitations due to emotional problems, and mental health. Participants self-report on items in a subscale that have between 2-6 choices per item using Likert-type responses (e.g. none of the time, some of the time, etc.). Summations of item scores of the same subscale give the subscale scores, which are transformed into a range from 0 to 100; 0= worst HRQL, 100=best HRQL. Higher scores indicate better health and well-being.
Change in ASAS response criteria | 6 weeks (at baseline and the end of follow-up)
  The Assessment in SpondyloArthritis international Society (ASAS) 20 response is defined as an improvement of >= 20% and absolute improvement of >= 1 unit (on a scale of 0 to 10) from Baseline in at least three of the following four domains, with no deterioration (where deterioration is defined as a worsening of >= 20% and a net worsening of >= 1 units [on a scale of 0 to 10]) in the remaining domains: Patient's Global Assessment, Pain, Function, Inflammation.
Change in pain, fatigue and stiffness by patient's Visual analogue scale (VAS) | 6 weeks (at baseline, 2-weeks, 4-weeks, end of follow-up)
  The VAS score assessed by participants, is used to determine the symptom (pain, fatigue and stiffness) impact due to AS in the past week. The level is measured in millimeters (mm) on a 100 mm horizontal line. The score ranges from 0 (no pain) to 100 (severe pain). Data are presented as mean VAS score +/- standard deviation.

SECONDARY OUTCOMES:
Individual evolution of intestinal Klebsiella | 6 weeks (at baseline, 2-weeks, 4-weeks, end of follow-up)
  To compare the average change of Klebsiella bacteria, quantified in colony-forming unit per gram of feces (cfu/gr) in faecal samples among each participant.
Change in Weight | 6 weeks (at baseline and the end of follow-up)
  To compare the average change in weight (kilograms) between LSD group and the controls, before and after the intervention.
Change in body mass index (BMI) | 6 weeks (at baseline and the end of follow-up)
  To compare the average change in BMI (kg/m2), calculated by weight/(height^2), between LSD group and the controls, before and after the intervention.
Change in body composition | 6 weeks (at baseline and the end of follow-up)
  To compare the average change in percentage of the evaluation of the body fat mass between LSD group and the controls, before and after the intervention.
Quantification of the average starch intake through 24h dietary recall | 6 weeks (3 days of each week till the end of follow-up)
  To quantify the average starch dietetic content (in grams per day), determined through the 24h dietetic recall applied for 3 days, to calculate the ingested starch during the intervention and determine the respective individual percentage of average reduction.

OTHER OUTCOMES:
Quantification of average dietetic starch | 5 days before baseline
  To quantify the usual individual daily dietetic intake of starch (grams per day), through the 24h dietary recall applied for 5 days.
Identification and quantification of intestinal microbiota | 6 weeks (at baseline and at the end of follow-up)
  To characterize the intestinal flora, namely, the presence of Klebsiella pneumoniae quantified in colony-forming unit per gram of feces (cfu/gr) in faecal samples.
Determination of height | at baseline
  To determine the height (meters) in all participants at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra MT Cardoso, MD, Principal Investigator — Universidade do Porto; Maria Leonor Silva, PhD, Study Director — Centro de Investigação Interdisciplinar Egas Moniz; Patrícia Padrão, PhD, Study Director — Universidade do Porto
Locations (1):
- Instituto Português de Reumatologia, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No